CLINICAL TRIAL: NCT02025777
Title: Evaluation of PillCam IBD Capsule Endoscopy System in Visualization of Lesions in the Colon Indicative of Ulcerative Colitis Disease
Acronym: UC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD-210
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; PillCam; IBD
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capsule endoscopy and colonoscopy (Experimental)
  Interventions: Device: Capsule Endoscopy

INTERVENTIONS:
Device: Capsule Endoscopy
  Other Names: CE

SUMMARY:
Study Hypothesis UC Disease affects the colon. PillCam IBD may be used for visualization of the colon mucosa in UC Disease patients. This study is designed to evaluate the yield and clinical impact of IBD capsule in detecting lesions associated with UC Disease and to determine the agreement between PillCam Platform with the IBD capsule and optical colonoscopy in the evaluation of UC disease extent.

Primary Scientific Objective To evaluate the agreement between PillCam IBD system and optical colonoscopy in the evaluation of UC disease extent (Non-active disease, Proctitis, Left-sided colitis, Pancolitis)

Proposed Design Established UC disease patients whose clinical condition suggests ongoing disease activity, aged 18 years and up, who have no evidence of symptomatic stricture or other obstruction that would prevent capsule passage will be enrolled in this study.

Patients will undergo bowel prep, followed by a PillCam IBD capsule examination and colonoscopy examination.

The Rapid videos will be evaluated by two readers, each from a different site, the colonoscopy videos will be evaluated by two other physicians, at the sites

INCLUSION CRITERIA

All subjects must fulfill all of the following inclusion criteria:

* Patients ages 18 years and up
* Patient has known UC according to physician discretion
* Patient has at least one positive inflammatory marker from the following:

  * ESR
  * CRP
  * CBC
* Patient is indicated and eligible for a standard of care colonoscopy examination
* Patient agrees to sign consent form

EXCLUSION CRITERIA

The presence of any of the following will exclude a patient from study enrollment:

* Crohn's Disease
* Antibiotic Associated Colitis
* Stool positive for O&P (C&S within 3 months of enrollment)
* Other known infectious cause of increased symptoms
* Known intestinal obstruction or current obstructive symptoms, such as severe abdominal pain with accompanying nausea or vomiting.
* Definite long stricture seen on radiological exam.
* Non-steroidal anti-inflammatory drugs including Aspirin, (twice weekly or more) during the 4 weeks preceding enrollment
* Suspected GI stricture, followed by patency capsule study or other imaging study that could not prove patency of the GI tract.
* Patient has had prior abdominal surgery of the gastrointestinal tract in the last 6 months, other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
* Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Patient with known gastrointestinal motility disorders.
* Subjects with known or suspected delayed gastric emptying
* Patient suffers from any condition, such as swallowing problems, which precludes compliance with study and/or device instructions.
* Patient has Type 1 or Type II Diabetes.
* Patient has any allergy or other known contraindication to the medications used in the study.
* Patient has any condition, which precludes compliance with study and/or device instructions.
* Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Concurrent participation in another clinical trial using any investigational drug or device.
* Patient suffers from a life threatening condition
* Patients with history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18 years and up
* Patient has known UC according to physician discretion
* Patient has symptoms of fresh bleeding and/or bloody diarrhea and/or at least one positive inflammatory marker within the past three months from the following:

  * ESR
  * CRP
  * CBC
* Patient is indicated and eligible for a standard of care colonoscopy examination for evaluation of disease activity and not for routine screening for dysplasia or colorectal cancer
* Patient agrees to sign consent form

Exclusion Criteria:

* Crohn's Disease
* Antibiotic Associated Colitis
* Stool positive for O&P and for C. difficile toxin within 3 months of enrollment
* Other known infectious cause of increased symptoms
* Known intestinal obstruction or current obstructive symptoms, such as severe abdominal pain with accompanying nausea or vomiting.
* Definite tight or long stricture seen on radiological exam.
* Non-steroidal anti-inflammatory drugs including Aspirin, (twice weekly or more) during the 4 weeks preceding enrollment
* Suspected GI stricture, followed by patency capsule study or other imaging study that could not prove patency of the GI tract.
* Patient has had prior abdominal surgery of the gastrointestinal tract in the last 6 months, other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
* Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Patient with a known gastrointestinal motility disorder.
* Subjects with known or suspected delayed gastric emptying
* Patient suffers from any condition, such as swallowing problems, which precludes compliance with study and/or device instructions.
* Patient has Type 1 or Type II Diabetes.
* Patient has any allergy or other known contraindication to the medications used in the study.
* Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Concurrent participation in another clinical trial using any investigational drug or device.
* Patient suffers from a life threatening condition
* Patients with history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Agreement between PillCam IBD system and optical colonoscopy in the evaluation of UC disease extent (Non-active disease, Proctitis, Left-sided colitis, Pancolitis) | 3 weeks post capsule procedure

SECONDARY OUTCOMES:
• Agreement between PillCam IBD system and optical colonoscopy in the evaluation of UC disease activity based on the Mayo Score (non-active, mild, moderate, severe) | 3 weeks after capsule procedure

OTHER OUTCOMES:
Type, incidence, severity, and duration of adverse events | 9 days after capsule procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yago González Lama, Dr., Principal Investigator
Locations (2):
- Sheari-Zedek Medical Center, Jerusalem, Israel
- Puerta de Hierro, Majadahonda, Madrid, Spain